CLINICAL TRIAL: NCT07229378
Title: Respiratory Muscle Strength Training to Prevent Dyspnea in the Newly Diagnosed Breast Cancer Patient Prior to Surgery"
Brief Title: Respiratory Muscle Strength Training to Prevent Respiratory Muscle Weakness in Adults Newly Diagnosed With Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB202501485
Record Dates: First submitted 2025-11-12; First posted 2025-11-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Respiratory muscle weakness; Breast Cancer; Breast Cancer Surgery; Respiratory strength training
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This research study is designed as a controlled, randomized, interventional trial for adults who have been diagnosed with breast cancer and are initiating breast cancer surgery. The feasibility, acceptability and strengthening effect of respiratory strength training exercises will be compared for effectiveness to a comparator group who will perform Guided Imagery exercises for at least ten sessions. This study design will examine which treatment is most beneficial in strengthening the respiratory musculature in preparation for breast cancer surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory muscle strength training (Experimental): Participants assigned to this arm will receive the equipment, education, and training to be able to perform respiratory muscle strength training for at least two weeks before breast cancer surgery.
  Interventions: Behavioral: Respiratory muscle strength training
- Guided Imagery Exercises (Active Comparator): Participants assigned to this group will receive education and training to be able to perform Guided Imagery, an exercise that uses relaxing, calming mental images, for at least two weeks prior to breast cancer surgery. This exercise does not provide respiratory strengthening and will thus be used as a comparator to respiratory muscle strength training.
  Interventions: Behavioral: Guided Imagery Exercises

INTERVENTIONS:
Behavioral: Respiratory muscle strength training — At the baseline visit, participants will receive an inspiratory muscle strength trainer pre-set for 40% of their measured maximal inspiratory pressure, and respiratory exercise education using a teach back method in the form of demonstration, as well as written instructions. The respiratory strength exercises are to be performed five days/week for at least two weeks, for a total of 45 breaths each day. Inspiratory respiratory muscle strength training for at least two weeks has been shown to reduce respiratory complications because of surgery in other populations (Lumb, 2019). Respiratory resistance will be increased by 10% each week following an assessment using the modified Borg scale, if participants rate the perceived level of exertion ≤ 5 (Mahler & Horowitz, 1994). Exercise diaries and weekly follow-up phone calls will be used to monitor and document exercises.
  Arms: Respiratory muscle strength training
Behavioral: Guided Imagery Exercises — Guided Imagery, a relaxation technique that utilizes visualization to develop relaxing, peaceful images to help improve emotional health by reducing anxiety, and stress. At the baseline visit, participants will receive training to perform Guided Imagery techniques using a teach back method in the form of demonstration and return demonstration for the exercise technique, as well as written instructions. Exercise diaries and weekly follow-up phone calls will be used to monitor and document exercises.
  Arms: Guided Imagery Exercises

SUMMARY:
The goal of this clinical trial is to learn if respiratory muscle strength training can prevent respiratory muscle weakness in adults who are newly diagnosed with breast cancer and are planning to have surgery. The main question it aims to answer is:

* Does respiratory muscle strength training in adults preparing for breast cancer surgery reduce the weakness that often occurs with surgery.

Researchers will compare Guided Imagery exercises to respiratory muscle strength training to see which is more helpful.

Participants will:

* Carry out respiratory muscle strength training or Guided Imagery exercises for at least 2 weeks at home.
* Meet with the researcher at home to complete breathing measurements before starting the exercises, after completing the exercises, and again after surgery.
* Keep a diary of the exercises that have been completed.

DETAILED DESCRIPTION:
Introduction and Challenge: The therapies required to treat breast cancer can cause side effects such as muscle weakness and breathing problems. Surgery, chemotherapy, radiation, and some necessary breast cancer drug treatments can all contribute to a weakness in breathing function. Additionally, respiratory muscle strength and flexibility decrease in older adults as a part of the natural aging process. Unfortunately, the combination of breast cancer treatments with aging can contribute to an increase in breathing problems. Weakened breathing muscles and less chest wall flexibility leads to a decreased ability to complete normal daily activities, potentially causing increased anxiety and depression, and an overall decrease in quality of life.

Respiratory muscle strength training is an exercise that has been found to specifically focus on building the muscle strength and function of breathing. Respiratory muscle strength training is an exercise that is performed while sitting in a chair at home, for 15 minutes each day. The participant inhales into a handheld device that provides resistance during inhalation. Respiratory muscle strength training has been successfully used in other people with chronic illnesses, lung cancer, cardiac surgery, head and neck cancer, and patients preparing for surgery. Recently, it was trialed in a group of breast cancer patients after surgery, combined with aerobic exercises, with reports that the group that received respiratory muscle strength training had better outcomes. However, respiratory strength training has not yet been used on its own, as a preventative exercise before breast cancer surgery.

Methods and Action Plan: In this proposed study, the investigators plan to compare a group of newly diagnosed breast cancer patients who carry out daily respiratory muscle strength training exercises, to a group of newly diagnosed breast cancer patients who perform daily Guided Imagery. Guided Imagery has been found to improve anxiety and depression through the use of relaxing mental images designed to activate the body-mind connection. The researcher will carry out the study visits and teaching in the participant's home. The study equipment is portable, and the daily exercises can be done at home. This will help reduce the newly diagnosed breast cancer patient's burden of participating in this study. The investigator will measure respiratory strength, breathing function, diaphragm muscle thickness, chest mobility, anxiety and depression, and quality of life before and after the respiratory muscle strength training and the Guided Imagery protocols, and compare the results of the two groups. Each participant will be taught how to perform the assigned exercises, filling out exercise diaries, and talking by phone with the researcher each week for progress updates about the exercises, as well as how difficult they feel the exercises are.

Results and Main Findings: The investigators hypothesize that the individuals who perform the respiratory muscle strength exercises will find the respiratory strengthening protocol acceptable, and will have stronger breathing muscles, better breathing function, more chest mobility, thicker diaphragms, less anxiety and depression, and increased quality of life scores than those who performed deep breathing exercises, and that the Guided Imagery group may experience less anxiety and depression. The investigators anticipate that older breast cancer patients will benefit more than younger breast cancer patients after performing respiratory strength training.

Conclusion and Impact: This study will provide the opportunity to test whether respiratory strength training is acceptable to newly diagnosed breast cancer patients, and whether it protects and supports the breast cancer patient from respiratory weakness prior to surgery. These results will also allow the investigators to assess the impact of respiratory strength training on the older breast cancer patient. If successful, the next steps will include developing a larger clinical trial to test a diverse population to ensure the protocol is successful, before integrating this exercise into standard clinical practice for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults (>18 years)
* Recently diagnosed with breast cancer
* Scheduled for breast cancer surgery
* English speaking, and can follow the protocol

Exclusion Criteria:

* Individuals who have already completed respiratory muscle strength training exercises
* Pregnancy,
* Recent pneumothorax
* Ruptured eardrum
* Uncontrolled hypertension, or uncontrolled reflux.
* Individuals who cannot complete at least ten exercise sessions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in maximal inspiratory pressure | Baseline, 2-4 weeks, and 2 weeks after surgery.
  Maximal inspiratory pressure (MIP) will be assessed as a measure of respiratory strength, using a respiratory pressure meter, a pocket-sized device that allows measures to be obtained with an accuracy of +/- 3%. Changes in MIP will be assessed at three timepoints.

SECONDARY OUTCOMES:
Change in Diaphragmatic thickness | Baseline, 2-4 weeks, and 2 weeks after surgery
  Diaphragm thickness will be measured with a handheld ultrasound device to record diaphragm thickness and at both end-inspiration and end expiration. A change in diaphragmatic thickness will be assessed at each of the three timepoints.
Change in Thoracic expansion | Baseline, 2-4 weeks, and 2 weeks after surgery.
  Thoracic expansion will be measured with a Gulick tape measure positioned around the participant's chest at the 4th intercostal space and will be used to record the difference between maximal inspiration and maximal expiration. The measures will be assessed at each of the three timepoints to assess for change over time.
Change in Dyspnea | Baseline, 2-4 weeks, and 2 weeks after surgery
  The Modified medical research council scale (MMRC) will be used to assess for a change in participants' dyspnea over the three timepoints. The MMRC scale includes a range of 0-4, with 4 being the most severe dyspnea.
Change in Anxiety and Depression | Baseline, 2-4 weeks, and 2 weeks after surgery.
  The Hospital Anxiety and Depression scale (HADS) is a two subscale, 14-question scale with Likert-style responses focused on feelings of anxiety and depression. A higher score represents increasing severity of symptoms of anxiety and/or depression. A change in scores will be assessed at each of the three timepoints.
European Organization for Research and Treatment of Cancer Core Questionnaire (EORTC QLQ-C30) | Baseline, 2-4 weeks, 2 weeks after surgery.
  The EORTC QLQ-C30 is a 30-item instrument developed to measure quality of life in cancer patients. Higher scores on the functional subscales indicate better functioning, while higher scores on symptom subscales describe higher symptom burden. A change in EORTC QLQ-C30 will be assessed at each timepoint.
Six Minute Walk Test Distance | Baseline, 2-4 weeks after the intervention, and 2 weeks after surgery.
  Standardized, functional capacity test by having the participant walk as far as possible on a flat, hard surface in six minutes.

OTHER OUTCOMES:
Feasibility and acceptability | Two weeks after surgery.
  Scores on a 6-question, Likert-style feasibility and acceptability questionnaire will be calculated, with higher scores indicating a higher participant perception of the feasibility and acceptability of the study.
Compliance with exercise diaries | Through study completion, an average of one year.
  Participant compliance with the exercise diaries will be assessed at the completion of the study and documented as a percentage. Higher scores will indicate stronger compliance.
Retention Rates | Through study completion, an average of one year.
  Retention rates will be reported at the completion of the study in the form of a percentage. Higher scores indicate a higher rate of participant retention.
Compliance with weekly phone calls | Through study completion, an average of one year.
  Compliance with weekly phone calls will be assessed at the end of the participant's study visits and reported as a percentage. Higher percentages indicate stronger compliance with phone calls

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K. Morgan, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that describe the results reported in this article, after the data is deidentified (tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following study publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee.

REFERENCES:
- [Background] Quinn CJ, Hydock DS. Effects of endurance exercise and doxorubicin on skeletal muscle myogenic regulatory factor expression. Muscles Ligaments Tendons J. 2018 Jan 10;7(3):418-425. doi: 10.11138/mltj/2017.7.3.418. eCollection 2017 Jul-Sep. PMID 29387634
- [Background] Nickels M, Erwin K, McMurray G, Talbot R, Strong M, Krishnan A, van Haren FMP, Bissett B. Feasibility, safety, and patient acceptability of electronic inspiratory muscle training in patients who require prolonged mechanical ventilation in the intensive care unit: A dual-centre observational study. Aust Crit Care. 2024 May;37(3):448-454. doi: 10.1016/j.aucc.2023.04.008. Epub 2023 Jun 14. PMID 37321882
- [Background] Nguyen BL, Baumfalk DR, Lapierre-Nguyen SS, Zhong R, Doerr V, Montalvo RN, Wei-LaPierre L, Smuder AJ. Effects of exercise and doxorubicin on acute diaphragm neuromuscular transmission failure. Exp Neurol. 2024 Aug;378:114818. doi: 10.1016/j.expneurol.2024.114818. Epub 2024 May 21. PMID 38782352
- [Background] Morton AB, Mor Huertas A, Hinkley JM, Ichinoseki-Sekine N, Christou DD, Smuder AJ. Mitochondrial accumulation of doxorubicin in cardiac and diaphragm muscle following exercise preconditioning. Mitochondrion. 2019 Mar;45:52-62. doi: 10.1016/j.mito.2018.02.005. Epub 2018 Feb 21. PMID 29474837
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Lumb AB. Pre-operative respiratory optimisation: an expert review. Anaesthesia. 2019 Jan;74 Suppl 1:43-48. doi: 10.1111/anae.14508. PMID 30604419
- [Background] Lovelace DL, McDaniel LR, Golden D. Long-Term Effects of Breast Cancer Surgery, Treatment, and Survivor Care. J Midwifery Womens Health. 2019 Nov;64(6):713-724. doi: 10.1111/jmwh.13012. Epub 2019 Jul 19. PMID 31322834
- [Background] Ibrahim AA, Gabr Ali AMM, Fadulelmulla IA, Ragab MMM, Aldemery AA, Mohamed AR, Dewir IM, Hakami HA, Hussein HM. Using Inspiratory Muscle Training to Improve Respiratory Strength, Functional Capacity, Fatigue, and Stress in Breast Cancer Patients Undergoing Surgery. J Multidiscip Healthc. 2024 May 1;17:1931-1941. doi: 10.2147/JMDH.S463961. eCollection 2024. PMID 38706507
- [Background] Gilliam LA, Moylan JS, Callahan LA, Sumandea MP, Reid MB. Doxorubicin causes diaphragm weakness in murine models of cancer chemotherapy. Muscle Nerve. 2011 Jan;43(1):94-102. doi: 10.1002/mus.21809. PMID 21171100
- [Background] Avudaiselvi T, Prabha SL. Effectiveness of Box Breathing Exercises in Reducing Stress among Women Postmastectomy: A Randomized Controlled Trial. J Pharm Bioallied Sci. 2025 Apr-Jun;17(2):75-77. doi: 10.4103/jpbs.jpbs_888_25. Epub 2025 Jul 23. PMID 40860007
- [Background] Al-Majid S, Wilson LD, Rakovski C, Coburn JW. Effects of exercise on biobehavioral outcomes of fatigue during cancer treatment: results of a feasibility study. Biol Res Nurs. 2015 Jan;17(1):40-8. doi: 10.1177/1099800414523489. Epub 2014 Feb 25. PMID 25504949